CLINICAL TRIAL: NCT01647620
Title: A Randomized, Double-blind, Placebo-controlled, Stepwise Study of the Pharmacokinetics (PK), Pharmacodynamics (PD), PK/PD Characteristics and Safety of Multiple Once-daily Oral Dosing of DPOC-4088 in Healthy Young Male Subjects
Brief Title: A Healthy Volunteer Study to Investigate the Blood Concentrations, the Effect on Blood Clotting and the Safety of Multiple Doses of DPOC-4088 Tablets in Different Doses.
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Diakron Pharmaceuticals couldn't fulfill the financial responsibility of the study
Sponsor: Diakron Pharmaceuticals (Industry)
Collaborators: University Ghent (Other); Kinesis Pharma B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DPOC-002
Record Dates: First submitted 2012-07-19; First posted 2012-07-23 (Estimated); Last update posted 2015-02-24 (Estimated); Status verified 2012-07

CONDITIONS: Deep Vein Thrombosis Leg; Stroke (in Patients With Atrial Fibrillation)
MeSH Terms: conditions — Venous Thrombosis; Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- DPOC-4088 (Active Comparator): A 10-day oral dosing of DPOC-4088 prolonged release tablet (20 hr release formulation). Starting dose in dose step 1 is 100 mg daily
  Interventions: Drug: DPOC-4088
- Placebo (Placebo Comparator): A 10-day oral dosing of matching placebo prolonged release tablet.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DPOC-4088 — A 10-day oral dosing of DPOC-4088 prolonged release tablet (20 hr release formulation). Starting dose in dose step 1 is 100 mg daily.
  Arms: DPOC-4088
Drug: Placebo — A 10-day oral dosing of matching placebo prolonged release tablet.
  Arms: Placebo

SUMMARY:
A study to investigate the concentrations of a new drug DPOC-4088 in blood, and to study the effect of this drug on blood clotting parameters. Furthermore the relation between the blood concentrations and the blood clotting effect will be investigated. Safety will be investigated as well. The objective of these investigations is to determine the optimal dose of DPOC-4088 that, achieves a relevant increase in a specific blood clotting parameter (the ecarin clotting time) without safety concerns.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, stepwise study of multiple once-daily oral dosing of DPOC-4088 (100 mg in Step 1) in healthy young male subjects. Each Step of the study will include 10 subjects and consist of screening for eligibility followed by a 13-day period during which once-daily oral doses of DPOC-4088 or placebo are administered for 10 consecutive days and blood is sampled for PK/PD measurements.

In each dose step, 8 subjects will receive active drug and 2 subjects will receive matching placebo according to a randomized allocation schedule.

During each Step, DPOC-4088 or placebo will be given each morning on Days 1 through 10, safety permitting. Each of the 10 days of dosing will be preceded by an overnight fast (10 hours). Subjects will have frequent PK/PD sampling performed for a 24 hour period following dosing on Day 1 and for a 72-hour period following dosing on Day 10. On Days 1 and 10, the first meal will be given at 4 hours post-dosing. On other dosing days, subjects will not have breakfast until one hour after dosing. Blood samples will be drawn for PK and PD evaluations immediately prior to dosing and at specified time intervals post-dosing. Following completion of all 10 days of dosing in each Step, subjects will return for a follow-up examination in 1 week (7-9 days).

After completion of all dosing in Step 1, PK, PD and safety data will be analyzed and (if necessary) used to determine the dose for Step 2, the same procedure will be followed for the next dose steps, if necessary.

The safety, tolerability, and the PK profile of DPOC-4088 will be assessed. Additionally, this study will assess the PD profile and the relationship of PK/PD in terms of the ability of DPOC-4088 to inhibit thrombin activity (based on prolongation of aPTT, ECT, TT and PT).

To main objective is to determine the dose of DPOC-4088 that, following multiple once-daily oral dosing, achieves a target increase of 2-fold over baseline in the ecarin clotting time (ECT) at the steady-state trough plasma concentration (Cmin-ss) without safety concerns.

ELIGIBILITY:
Inclusion Criteria:

1. Male between 18 to 50 years of age inclusive.
2. Either a non- or a light-smoker (<5 cigarettes per day) and agrees to refrain from smoking from the evening prior to first dosing until after the last PK sample of each step is drawn.
3. Body-mass index (BMI) of 18-32 kg/m2.
4. In good health on the basis of history, physical examination, and routine laboratory data.
5. Understands the procedures and agrees to participate in the study program by giving written informed consent.
6. Coagulation tests including aPTT, ECT, TT and PT within the reference range and a platelet count >145,000/mm3.
7. At screening, normal transaminases and negative Hemoccult Sensa(R) test. In the event of a positive Hemoccult test, the test should be repeated twice. If the results of both repeats tests are negative, the first Hemoccult test result is considered a false positive and the subject may be included.

Exclusion Criteria:

1. Mentally or legally incapacitated, significant emotional problems at the time of the study, or a history of psychiatric disorders within the last 10 years.
2. History within the last 10 years of asthma or other pulmonary disease, major cardiovascular, hepatic, endocrine (including diabetes), rheumatological, or renal disease or of prior spine or disc surgery.
3. History within the last 10 years of neurologic disease including stroke, transient ischemic attacks, seizure, head trauma, neurological tumors, brain or spinal cord surgery, neuropathy, or neuromuscular illness.
4. Active gastrointestinal disease including: peptic ulcer disease, gastritis, clinically significant Helicobacter pylori infection, inflammatory bowel disease, diverticular disease, colonic polyps, or of any gastrointestinal malignancy, or recent (within 3 weeks) benign enteritis.
5. History of any illness or condition that, in the opinion of the investigator, might confound the results of the study or pose additional risk in administering study drug to the subject (e.g., surgery within the previous 3 months).
6. Donated a unit of blood (450 mL) or participated in another clinical study drug trial within the 4 weeks prior to screening.
7. Family or personal history of bleeding disorders, including von Willebrand's disease.
8. History of significant gingivitis or other periodontal disease.
9. Received any prescription anticoagulant within the 30 days preceding screening including but not limited to warfarin, heparin, low-molecular weight heparin, hirulog, hirudin, argatroban, or dabigatran.
10. Has received 14 days prior to first dosing or anticipates needing during the study any prescription or nonprescription (including over the counter) preparation that contains aspirin (including low-dose aspirin), ibuprofen, indomethacin, diclofenac, naproxen, meloxicam, any other NSAID or NSAID-containing product such as pain relievers, cold or sinus remedies, or any other drug which influences platelet aggregation.
11. Received any investigational drug within the 30 days preceding screening.
12. Regular user of any medication (including over-the-counter medication) for 14 days prior to first dosing, except for acetaminophen. Subject currently uses prescription or nonprescription drugs on a regular basis which cannot be discontinued for 14 days prior to first dosing until the last study visit (including "recreational use" of illicit drugs). Subject has a recent history (within the last 2 years) of drug or alcohol abuse.
13. Subjects unable to stop using the following medications during the study (from first dosing until after the last study visit): erythromycin or erythromycin-like drugs, clarithromycin, diltiazem, cimetidine, warfarin-like anticoagulants, cyclosporine, itraconazole (or other systemic antifungal agents in the azole class), nefazodone, selective serotonin reuptake inhibitors (SSRI antidepressants), benzodiazepines, any systemic immunosuppressive agents (including glucocorticoids), cisapride and the H1 antagonists terfenadine and astemizole, and HIV protease inhibitors.
14. Unable to refrain from the use of antacids, H2 blockers, sucralfate, or proton pump inhibitors beginning 14 days prior to first dosing until the last study visit.
15. Has had major surgery within previous 3 months prior to first dosing or is anticipated to have major surgery within 2 weeks after completion of the study.
16. Positive hepatitis serology (HBsAg and anti-HCV) showing any sign of active hepatitis.
17. History of any chronic and/or active hepatic disease including hepatitis or biliary tract disease. Any subject with a history of hepatitis B or C at screening will be excluded. Subjects with a history of self-limited hepatitis A with complete resolutions documented at ≥12 months prior to entry would be eligible for inclusion.
18. HIV positive.
19. Significant unexplained and/or reproducible abnormalities on pre-study clinical examination or laboratory measurements.
20. History of significant drug allergy or any clinically significant adverse event of a serious nature related to the administration of either a marketed or investigational drug.
21. Known history of fainting from phlebotomy or from minor trauma resulting in bleeding.
22. Habitual heavy consumer of coffee (more than 6 cups of coffee/day).
23. Unable to refrain from consumption of grapefruit or grapefruit juice for at least 14 days prior to first dosing until the last study visit.
24. Unable to refrain from the use of St. Johns wort for at least 14 days prior to first dosing until the last study visit.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-02; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
The dose of DPOC-4088 that, following multiple once-daily oral dosing, achieves a target increase of 2-fold over baseline in the ecarin clotting time (ECT) at the steady-state trough plasma concentration (Cmin-ss) without safety concerns

SECONDARY OUTCOMES:
The dose of DPOC-4088 that, following multiple once-daily oral dosing, achieves a target increase of 1.5-fold over baseline in the activated partial thromboplastin time (aPTT) at Cmin-ss without safety concerns.
The extent and duration (at the end of dosing) of inhibition of coagulation parameters as measured by the change from baseline in ECT and aPTT.
The DPOC-4088 plasma concentration vs time profile and Cmax-ss/Cmin-ss following multiple once-daily oral dosing.
The safety of DPOC-4088 given once-daily for 10 days.
  Vital sign measurements, 12-lead ECGs, physical examinations, laboratory and adverse events.
  A complete physical examination and a brief neurological examination will be performed pre-study and post-study. On Days 2, 4, 5, 7, and 10, the physical examination is limited to examination of the skin for evidence of bleeding, bruising or petechiae.

CONTACTS AND LOCATIONS:
Overall Officials: Luc M van Bortel, Prof. Dr., Principal Investigator — University Ghent
Locations (1):
- Drug Research Unit Ghent, Ghent, Belgium